CLINICAL TRIAL: NCT01076907
Title: Can Simple and Inexpensive Techniques Enhance Patient Comfort in Sedation-risk Free Screening and Surveillance Colonoscopy?
Brief Title: Techniques to Enhance Patient Comfort in Sedation-risk Free Colonoscopy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Necessary equipment to perform the study arms was removed by the medical center administration.
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Felix W. Leung, Staff Physician, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FL0055
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Screening of Colonic Polyps
Keywords: colonoscopy; polyps
MeSH Terms: conditions — Polyps | interventions — Air

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warm water loading of sigmoid colon (Experimental): Warm water loading of sigmoid colon and irrigation when spasms occur.
  Interventions: Other: Warm water
- Control (Placebo Comparator): No water loading, only air and waiting for spasms to subside.
  Interventions: Other: Control

INTERVENTIONS:
Other: Warm water — Warm water loading of sigmoid colon when spasms occur and waiting for them to subside.
  Arms: Warm water loading of sigmoid colon
Other: Control — Air will be used instead of warm water for unsedated colonoscopy.
  Other Names: air
  Arms: Control

SUMMARY:
Hypotheses

1. Loading the sigmoid colon with warm water and warm water irrigation for dealing with spasm (Study Treatment) will significantly reduce the proportion of patients complaining of abdominal discomfort compared with no water loading and waiting for spasms to subside (Control Treatment). The median discomfort score reported by the patients will be significantly lower in the group receiving the Study Treatment than the group receiving Control Treatment. Hypothesis
2. Exploratory hypothesis: There are differences in secondary outcome variables when patients managed by the Study and Control Treatments are compared. Co-variables affect the primary and secondary outcome variables.

DETAILED DESCRIPTION:
The purpose of the study is to conduct a RCT study to determine the effectiveness of loading the sigmoid colon with warm water and warm water irrigation for dealing with colonic spasms in enhancing patient abdominal comfort during unsedated colonoscopy. The specific aim is to compare Study Treatment of warm water loading and irrigation when spasms occur with Control Treatment of no water loading and waiting for spasms to subside. The proportion of patients complaining of abdominal discomfort and their discomfort score are the primary outcome variables. The secondary outcome variables and co-variables described below will be recorded in a prospective manner to ensure completeness of data collection. In preliminary clinical observation at VA Sepulveda ACC, 25 to 30% of VA patients accept colonoscopy without sedation. The goal of this study is to find ways of further reducing discomfort associated with unsedated colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Accepts adult healthy male and female patients
* At least 18 years of age
* In need of colonoscopy for screening or follow up of colonic polyps
* Willing to consent and be randomized

Exclusion Criteria:

* Patients receiving outpatient narcotic treatment
* Patients who report excessive anxiety
* Patients with moderate to severe abdominal discomfort
* Unable to provide consent
* Have poor bowel preparation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
abdominal discomfort | 30 days
  Abdominal discomfort reported to a blinded observer 5-10 min after colonoscopy.

SECONDARY OUTCOMES:
colonoscopy-related outcomes | 30 days
  various procedure related measures

CONTACTS AND LOCATIONS:
Overall Officials: Felix W. Leung, MD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (1):
- Greater Los Angeles Healthcare System and the Sepulveda Ambulatory Care Center, Los Angeles, California, United States